CLINICAL TRIAL: NCT01039090
Title: Prospective, Randomised, Comparative Study Comparing Efficacy of Continuous Apomorphine Infusion Versus Usual Dopaminergic Per os Treatment on Cognitive and Neuropsychological Functions in Parkinson's Disease: a Clinical and PET-scan Study
Brief Title: Efficacy of Continuous Apomorphine Infusion on Cognitive and Neuropsychological Functions in Parkinson's Disease
Acronym: APO-TEP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-006045-10; LOC/08-08
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Parkinsons's Disease
Keywords: Not eligible for deep brain stimulation; Parkinsons's patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Per os dopaminergic treatment (Active Comparator)
  Interventions: Drug: Usual dopaminergic per os treatment
- Continuous Apomorphine infusion (Experimental)
  Interventions: Drug: Continuous Apomorphine infusion

INTERVENTIONS:
Drug: Continuous Apomorphine infusion — Continuous Apomorphine infusion during 6 months
  Arms: Continuous Apomorphine infusion
Drug: Usual dopaminergic per os treatment — No specific change in the dopaminergic per os treatment
  Arms: Per os dopaminergic treatment

SUMMARY:
In Parkinson's disease, treatment mainly aims to improve motor functions. However, other dysfunctions are often observed in Parkinson's patients, and may have important consequences on the quality of life of patients.

Cognitive and neuropsychological troubles may be observed, as memory impairment or anxiety for example. As this kind of troubles is worrying for the patient himself (herself) and his/her family, treatment needs to take into account those troubles in addition to motor difficulties. In our centre, we have already used continuous Apomorphine infusions among Parkinson's patients and it seems to have good results. The present study aims to objectively assess the efficacy of continuous Apomorphine infusions on cognitive and neuropsychological functions in Parkinson's disease using clinical and positron emission tomography (PET)-scan measures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and more
* Parkinson's disease according to UKPDSBB diagnosis criteria
* Motor difficulties in spite of dopaminergic per os treatment
* Not eligible for deep brain stimulation for one or more reasons (age>70, axial troubles in spite of dopaminergic per os treatment, cognitive troubles and/or hallucinations)

Exclusion Criteria:

* Mattis scale < 120
* Contraindication to Apomorphine (liver insufficiency, severe cognitive troubles, allergy, pregnancy, neuroleptic treatment)
* Contraindication to Fluoro-Deoxy-Glucose which is used in PET-Scan (allergy, kidney failure, pregnancy, breast feeding)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Neuropsychological results: Montgomery-Åsberg Depression Rating Scale (MADRS), The Lille Apathy Rating Scale (LARS), Spielberger | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc VERIN, MD PhD, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France

REFERENCES:
- [Result] Auffret M, Le Jeune F, Maurus A, Drapier S, Houvenaghel JF, Robert GH, Sauleau P, Verin M. Apomorphine pump in advanced Parkinson's disease: Effects on motor and nonmotor symptoms with brain metabolism correlations. J Neurol Sci. 2017 Jan 15;372:279-287. doi: 10.1016/j.jns.2016.11.080. Epub 2016 Dec 2. PMID 28017228